CLINICAL TRIAL: NCT00574236
Title: A Phase II Trial of Bortezomib and Doxorubicin in Metastatic Breast Cancer
Brief Title: Phase II Trial of Bortezomib and Doxorubicin in Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: no additional funding
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0130; CO04101; A534260 (Other: UW Madison); SMPH/MEDICINE (Other: UW Madison)
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Results first posted 2018-04-20 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2018-04

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bortezomib; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Drug: PS-341, doxorubicin

INTERVENTIONS:
Drug: PS-341, doxorubicin — bortezomib:1.3 mg/m2 IVP over 3-5 sec. days 1, 4, 8, 11 of 21 day cycle doxorubicin: 20 mg/m2 IV over 3-5 min. days 1,8 (one hour after bortezomib) of 21 day cycle
  Other Names: Velcade; Adriamycin

SUMMARY:
Primary objective is to determine the effectiveness of the combination of bortezomib and doxorubicin in patients with metastatic breast cancer. The trial format is a single arm Phase II design wherein patients are treated with bortezomib IV on days 1, 4, 8, and 11 and with doxorubicin IV on days 1 and 8 of a 21-day cycle.

ELIGIBILITY:
Inclusion Criteria:

* Cytologically or histologically confirmed metastatic breast cancer
* Measurable or evaluable disease
* Age > 18, PS 0,1,2
* MUGA > 45%
* Received one or fewer chemotherapies or investigational regimens for metastatic disease, no limit to the number of prior hormonal therapies. May have had single agent Herceptin and/or Herceptin plus single-agent chemotx.
* Must meet designated laboratory criteria within 14 days of enrollment

Exclusion Criteria:

* Doxorubicin for metatstatic disease.
* Pregnant or lactating.
* Active infections, no myocardial infarction within 2 months of enrollment.
* Investigational drugs within 14 days of enrollment.
* Chemotherapy, radiotherapy, hormonal therapy or other investigational therapy within 4 weeks of enrollment.
* Neuropathy that is > grade 2.
* Active brain mets.
* Hypersensitivity to bortezomib, boron, or mannitol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-08 (Actual); Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Stewart, M.D., Principal Investigator — University of Wisconsin PPC Comprehensive Cancer Center
Locations (1):
- University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled subjects with metastatic breast cancer from the Wisconsin Oncology Network (WON), which is driven by investigators at the University of Wisconsin Carbone Cancer Center, from August of 2006 through February of 2008.
Groups:
- Bortezomib and Doxorubicin: Subjects received therapy on days 1, 4, 8, and 11 of a 21-day cycle. 1.3 mg/m2 of Bortezomib was administered intravenously over 3-5 seconds on days 1, 4, 8, and 11, no less than 72 hours apart. 20 mg/m2 of Doxorubicin was administered intravenously over 3-5 minutes on days 1 and 8, one hour after Bortezomib administrations.
Period: Overall Study
Arm/Group | Bortezomib and Doxorubicin
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Bortezomib and Doxorubicin
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Determine the clinical efficacy of bortezomib and doxorubicin in patients with metastatic breast cancer. Overall response rate is defined as both complete and partial response per RECIST, where complete response is the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm. Partial response is defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive disease is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5mm.
Time Frame: Every two cycles/42 days, up to 7 months
Population: Protocol accrued only 4 of 54 subjects, and was ultimately terminated. No data analysis was done.
Measure: Count of Participants; unit: Participants
Arm/Group | Bortezomib and Doxorubicin
Number analyzed (Participants) | 4
Participants
  Complete Response | 0
  Partial Response | 1
  Progressive Disease | 3

2. Secondary Outcome: Time to Progression
Description: Number of days to progression, where progression is defined as the number of days from the day of first study drug administration to the day the patient experiences an event of disease progression, or the appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. If a patient has not experienced an event of disease progression, then the patient's data will be censored at the date of the last available evaluation. Progression-free survival will be summarized by medium time to progression.
Time Frame: Up to one year
Measure: Median (Full Range); unit: days to progression
Arm/Group | Bortezomib and Doxorubicin
Number analyzed (Participants) | 4
days to progression | 47 [41 to 210]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 1 year, 9 months.
Description: Investigators conducted continuous reviews of data and participant safety at monthly meetings, where the results of each of each participant's treatment were discussed and the discussion was documented in the minutes.
Arm/Group | Bortezomib and Doxorubicin
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bortezomib and Doxorubicin (N=4)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 4 (5)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 (5)
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 1 (1)
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 3 (3)
Heartburn/dyspepsia (Gastrointestinal disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (2)
Infection with normal ANC or Grade 1 or 2 neutrophils - Ungual (nails) (Infections and infestations) | 1 (1)
Infection with normal ANC or Grade 1 or 2 neutrophils - Vagina (Infections and infestations) | 1 (1)
Insomnia (General disorders) | 1 (1)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1)
Mood alteration: Depression (Nervous system disorders) | 1 (1)
Mucositis/stomatitis (functional/symptomatic) - Oral cavity (Gastrointestinal disorders) | 1 (2)
Nail changes (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (6)
Neuropathy: cranial - CN V Motor-jaw muscles; Sensory-facial (Nervous system disorders) | 1 (1)
Neuropathy: sensory (Nervous system disorders) | 3 (5)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 2 (2)
Pain (General disorders) | 4 (9)
Sweating (diaphoresis) (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No